CLINICAL TRIAL: NCT06389851
Title: Evaluation of the Effects of Tomato Consumption on the Parameters of Hepatic Steatosis, Intestinal Function and on Glucose and Lipid Metabolism in Subjects With NAFLD
Brief Title: Effects of Tomato Consumption on Steatosis, Intestinal Function and Glucose and Lipid Metabolism in Subjects With NAFLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Dr. Di Stasi Vincenza (Unknown); Dr. Donvito Rosanna (Unknown); Dr. Cozzolongo Raffaele (Unknown); Dr. Giannuzzi Vito (Unknown); Dr. Zappimbulso Marianna (Unknown); Dr. Shahini Endrit (Unknown); Dr. Notarnicola Maria (Unknown); Dr. Russo Francesco (Unknown); Dr. Riezzo Giuseppe (Unknown); Dr. Donghia Rossella (Unknown); Dr. Cesternino Anna Maria (Unknown); Dr. Cici Rosalisa (Unknown); Dr. Cerabino Nicole (Unknown); Dr. Martina Di Chito (Unknown); Dr. Pesole Pasqua Letizia (Unknown); Dr. Coletta Sergio (Unknown); Dr. Stabile Dolores (Unknown); Dr. Ancona Anna (Unknown); Dr. D'Attoma Benedetta (Unknown); Dr. Ignazzi Antonia (Unknown); Dr. De Nunzio Valentina (Unknown); Dr. Tatoli Rossella (Unknown); Dr. Pinto Giuliano (Unknown)
Responsible Party: Principal Investigator, Prof. Giovanni De Pergola, MD, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD-LYCOPENE
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: NAFLD; IBS
Keywords: NAFLD; Liver Diseases; IBS
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Intervention Model Description: The study evaluates the effects on NAFLD, Intestinal Integrity and Microbiota of a diet enriched with tomatoes compared to a diet without tomatoes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Group - Tomato-free diet (Experimental): Subjects assigned to this arm will follow a tomato-free diet
  Interventions: Dietary Supplement: Experimental: Case Group - Tomato-free diet
- Case group - Diet enriched with tomatoes (Experimental): Subjects assigned to this group will follow a diet with pre-established quantities of tomato and sauce
  Interventions: Dietary Supplement: Experimental: Case group - Diet enriched with tomatoes

INTERVENTIONS:
Dietary Supplement: Experimental: Case Group - Tomato-free diet — Nutritional intervention without tomatoes and sauce
  Other Names: Tomato-free diet
  Arms: Case Group - Tomato-free diet
Dietary Supplement: Experimental: Case group - Diet enriched with tomatoes — Nutritional intervention enriched with tomatoes and souce
  Other Names: Diet enriched with tomatoes
  Arms: Case group - Diet enriched with tomatoes

SUMMARY:
The study in question is an interventional study with nutritional intervention. the aim of the study is to evaluate whether a diet enriched with tomatoes can have favorable effects on:

* specific aspects associated with NAFLD, such as the degree of hepatic steatosis and fibrosis;
* circulating levels of molecules correlated with the degree of generalized and hepatic inflammation and the blood concentrations of metabolic and cardiovascular risk factors associated with abdominal obesity;
* intestinal barrier;
* body composition;
* intestinal microbiota;
* symptoms of IBS (irritable bowel syndrome) in patients with NAFLD.

DETAILED DESCRIPTION:
Chronic liver diseases are among the leading causes of morbidity, mortality. The increase in mortality from liver disease has been associated with the greater prevalence of NAFLD, which is, the most frequent chronic liver disease observed in clinical practice in Western countries. The term "hepatic steatosis" is the hallmark of NAFLD and refers to a fat deposit in the liver cells greater than 5% and which is not related to alcohol intake or viral infections or the use of drugs. It is possible to distinguish between hepatic steatosis and non-alcoholic steatohepatitis (NASH), a subtype of NAFLD in which fat deposition is associated with lobular inflammation, with or without fibrosis, characterized by the risk of possible progression to liver cirrhosis and, possibly, to hepatocellular carcinoma. Hepatic steatosis is an independent risk factor for all liver alterations that characterize NAFLD, particularly inflammation and fibrosis. Globally, the prevalence of NAFLD, assessed by liver ultrasound, is on average 30.69%. In the last 10-15 years its prevalence, always assessed by liver ultrasound, has increased by +38.7%, going from 25.16% in the period 1990-2006 to 34.59% in the period 2016 -2019. If the highest prevalence of NAFLD is in Latin America (44.37%), it is 31.2% in North America and 25.1% in Western Europe. Studies conducted in Italy indicate a prevalence of NAFLD of 22.5 -27.0% in the general population, with a 2 % prevalence of fibrosis, diagnosed by non-invasive means. In patients with NAFLD, the mortality rate for all causes is equal to 12.60 per 1000 person-years, while that from cardiovascular causes, extra-hepatic tumors and liver-related causes is, respectively, equal to 4.20 per 1000 people/year,2.83 per 1000 person-years and 0.92 per 1000 person-years. In the onset and progression of NAFLD, alongside the role of insulin resistance and generalized inflammation, pathways of relationship between the intestine and the liver are also involved, in turn influenced by the type of intestinal microbiota. Age also influences the evolution of these liver diseases and, as they advance, the prevalence of NAFLD and related fibrosis increases. Furthermore, the prevalence of NAFLD increases in parallel with the increase in the presence of metabolic alterations such as dyslipidemia and type 2 diabetes mellitus. Al though the main causes of death in people affected by NAFLD are cardiovascular diseases and extrahepatic malignancies, fibrosis hepatic advanced appears to be "in itself" an unfavorable prognostic marker for the outcomes of liver diseases. In the absence of officially approved pharmacological therapies for the treatment of NAFLD, European clinical guidelines and systematic reviews with meta-analyses recommend lifestyle-based interventions. These mainly involve quantitative and qualitative changes in diet and an increase in regular physical exercise, considered together as the best therapeutic strategy for the management of patients with NAFLD. Diet can improve NAFLD by reducing the amount of liver fat and insulin resistance, while exercise promotes weight loss and improves liver function. The diet therefore acts as an effective prevention tool in combating metabolic-related diseases, such as NAFLD. In particular, fruit with its high content of polyphenols has been shown to exert a high anti-inflammatory, antithrombotic and antiproliferative action. Recently, it has been demonstrated in vitro on human colorectal carcinoma cell lines that table grape polyphenolic extracts can inhibit cell proliferation and growth as well as influence the morphology of the cell, inhibiting its migration capacity. These data support the idea that grapes, as a nutraceutical, can have health effects and prevent the mechanisms of oxidation, cellular inflammation and metastasis. Furthermore, a clinical trial on healthy volunteers demonstrated that the daily intake of grapes can down-regulate the expression of small single-stranded non-coding RNA molecules, called miRNAs, metabolically associated with the "metabolism of cancer of the gastrointestinal tract". Therefore, their inhibition would lead to preventing the transformation of the cell in a neoplastic sense. Recently, among food antioxidants, particular attention has been paid to lycopene, a phytochemical belonging to the carotenoid family. Lycopene is found abundantly in vegetables and is responsible for their characteristic color. Its bioactive properties are influenced by many factors, such as bioavailability, metabolism and interaction with other carotenoids. In nature, lycopene occurs in its trans isoform, which is responsible for its bioavailability in the presence of elevated temperatures (trans to cis). It is assumed that due to the cis form, lycopene is more highly bioavailable. Since it is a fat-soluble substance, the associated consumption of dietary fats amplifies its bioavailability. The main sources of lycopene in the Mediterranean diet are tomatoes and tomato products. In the European population, lycopene consumption varies between 5 and 7 mg/day and over 80% of its daily intake comes from tomato-based products. Several studies have demonstrated the beneficial effects of lycopene on health resulting from its structure and lipophilic nature, which determines its anti-inflammatory and antioxidant effects. Recent studies suggest that changes in the intestinal microbiota may represent a new strategy to prevent or treat NAFLD and it is now known that a specific diet and regular physical exercise can induce changes in the composition of the intestinal microbiota, which in turn contribute to an increase of insulin. sensitivity and hepatic lipid metabolism. Furthermore, a recent prospective study observed that NAFLD is associated with an increase in 20% risk of developing irritable bowel syndrome (IBS), a disease not due to organic lesions and characterized by abdominal pain and abdominal swelling, associated with frequent diarrhea or prolonged constipation, often in periodic alternation, relief of symptoms after defecation, modification of the frequency of bowel movements and/or consistency of the stool. IBS affects 4.1% to 10.1% of the general population and is responsible for a reduction in the quality of life and an increase in healthcare costs and, therefore, it is a priority to identify lifestyle factors that can improve the IBS symptoms.Since NAFLD and IBS share variations in circulating levels of proinflammatory cytokines(increased tumor necrosis factor (TNF)-α, interleukin (IL)-6, etc and reduction in IL-10),cross-talk between the liver- brain-gut and gut-liver axis, dysfunction of the intestinal microbiota, alterations of the intestinal barrier and alterations of intestinal motility, it cannot be excluded that the improvement or worsening of NAFLD may favor the improvement or worsening of IBS. Furthermore, it has been seen that the mechanisms that regulate intestinal barrier function are altered in NAFLD and this situation represents an aggravating factor. Inflammation associated with liver disease may in turn play a significant role in the development of gastrointestinal (GI) disorders. It is a chronic low intensity state that involves the entire organism. Inflammation is related to an increase in inflammatory cytokines in tissues which,by activating immune responses, alter cellular metabolic pathways. In general, chronic low-level inflammation and the variation in the concentration of metabolic hormones, together with the distribution of adipose tissue in the abdominal cavity and alterations in the bacterial populations of the intestinal microbiota, represent the main factors involved in the development of gastrointestinal pathologies that they develop precisely through alterations of the intestinal barrier. The intestinal barrier can be considered a dynamic system that also responds to humoral signals and to a series of different molecules which, in various ways, are called into question. Among these, it is important to consider zonulin, a GI peptide capable of modulating the functionality of tight junctions (TJs). Serum zonulin levels have been shown to correlate with the extent of mucosal barrier impairment. Cellular and/or TJ damage can have a significant impact on the correct function of intestinal permeability (PI). The I-FABPs (intestinal fatty acid binding proteins) are cytosolic proteins present in epithelial cells responsible for the transport of fatty acids. They can be released into the circulation following the loss of membrane integrity and are rapidly eliminated in the urine; therefore, they represent non-invasive markers of early damage at the cellular level of the intestinal epithelium. Likewise the heck oxidase (DAO), an intracellular enzyme with a high level of activity in the upper layer of the intestinal villi, is considered a serum marker of intestinal epithelial integrity. Alterations in the barrier function can favor the entry of bacteria and their products. Lipopolysaccharide (LPS), a predominant component in the cell wall of Gram-negative bacteria, has been found to influence barrier function. Under physiological conditions, LPS is unable to cross intact epithelium, but in the presence of reduced epithelial integrity, it can cross the GI barrier. Tryptophan is an essential amino acid for humans since it is not synthesized in humans; commensal bacteria catabolize tryptophan into various derivatives, which are absorbed by the intestine and eliminated in the urine. Two of these compounds, indoxyl sulfate and 3-methyl-indole (skatole), are currently used to diagnose small intestinal and colon dysbiosis.

The study will be a randomized and controlled study with nutritional intervention: 60 subjects, suffering from NAFLD, will be enrolled and randomly assigned to the two groups of the study:

Group A (Treatment): the subjects enrolled in this group will have to consume 200g of fresh raw tomatoes and 50g of sauce per day Group B (Control): the subjects enrolled in this group must comply with one diet free of tomatoes All groups will be provided with instructions on the diet to follow, depending on the arm to which they will be assigned. The treatment will last 6 weeks and, in addition to the V0 (Screening Visit), 2 other visits (V1-V2) are planned.

At V0, will be subjected to: Medical history; Fibroscan, to evaluate the degree of NAFLD; - Detection of anthropometric characteristics; BIA Test.

Enrolled patients will be invited to return for V1, after 7 days to receive the personalized diet. In V1, they will be subjected to blood sampling and body composition assessment using DEXA. Whole blood and serum samples will be used for the measurement of routine blood chemistry parameters and nutritional, metabolic and cardiovascular risk parameters. The HOMA index and the degree of hepatic steatosis FLI and FIB-4 will be calculated. The main adipokines (leptin, RBP-4, visfatin), the main hepatic growth factors (HGF, Fetuin-A, FGF21, FGF19, PAI-1) and the main proinflammatory cytokines (highly sensitive C-reactive protein, IL-6 , IL-8, TNF-α) and anti-inflammatory (IL-4); other aliquots will be used for lipidomics and biochemical analyses. On the serum samples taken from the subjects at times V1 and V2, the antioxidant activity and the inflammatory state and the serum levels of the deglycant enzymes will be evaluated, through the study of the SOD1 and SOD2 enzymes, IL-6, TNF-alpha and the Fructosamine 3-Kinase and glyoxalase. The study subjects will also be asked to bring two stool samples for the evaluation of the intestinal microbiota and for the measurement of fecal Zonulin and the fecal metabolome, as well as two urine samples.

Optional visits Patients enrolled in the study will be asked, on an optional and voluntary basis, to undergo two outpatient sigmoidoscopies with cold biopsies if they wish to undergo.

A sigmoidoscopy after the screening visit, the second would be performed at the end of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI≤30;
* Diagnosis of hepatic steatosis, formulated on the basis of criteria

Exclusion Criteria:

* Patients with BMI > 30;
* Presence of any pathology that could influence the presence of steatosis apart from the pathologies that represent inclusion criteria;
* Pregnancy or breastfeeding;
* Serious medical conditions that may compromise participation in the trial;
* People following a special diet.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
The effect of intervention on CAP value (Controlled Attenuation Parameter) | at Baseline and after 6 days weeks
  To evaluate whether the adoption of a diet enriched with tomato and sauce in patients suffering from NAFLD can exert favorable effects, after 6 weeks of treatment, on the CAP value (Controlled Attenuation Parameter), a parameter which evaluates the level of Liver Fibrosis, measured by Fibroscan.
The effect of intervention on FLI value (fatty liver index) | at Baseline and after 6 days weeks
  To evaluate whether the adoption of a diet enriched with tomato and sauce in patients with NAFLD can exert favorable effects on the FLI value (fatty liver index), based on anthropometric parameters (BMI, abdominal circumference) and blood chemistry (triglycerides and γGT)
The effect of intervention on routine blood chemistry parameters, relating to NAFLD and fibrosis | at Baseline and after 6 days weeks
  To evaluate whether the adoption of a diet enriched with tomato and sauce in patients with NAFLD affects routine blood chemistry parameters. The following will be taken into consideration: Blood sugar, Glycated hemoglobin, triglycerides, total cholesterol
The effect of the intervention on the integrity of the intestinal barrier | at Baseline and after 6 days weeks
  To evaluate whether the adoption of a diet enriched with tomato and sauce in patients with NAFLD affects the integrity of the intestinal barrier and the microbiota
The effect of the intervention on the microbiota | at Baseline and after 6 days weeks
  To evaluate whether the adoption of a diet enriched with tomato and sauce in patients with NAFLD affects the microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Saverio de Bellis, Castellana Grotte, BARI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younossi ZM, Golabi P, Paik JM, Henry A, Van Dongen C, Henry L. The global epidemiology of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH): a systematic review. Hepatology. 2023 Apr 1;77(4):1335-1347. doi: 10.1097/HEP.0000000000000004. Epub 2023 Jan 3. PMID 36626630
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Saini RK, A Bekhit AE, Roohinejad S, Rengasamy KRR, Keum YS. Chemical Stability of Lycopene in Processed Products: A Review of the Effects of Processing Methods and Modern Preservation Strategies. J Agric Food Chem. 2020 Jan 22;68(3):712-726. doi: 10.1021/acs.jafc.9b06669. Epub 2020 Jan 7. PMID 31891495
- [Background] Wu S, Yuan C, Yang Z, Liu S, Zhang Q, Zhang S, Zhu S. Non-alcoholic fatty liver is associated with increased risk of irritable bowel syndrome: a prospective cohort study. BMC Med. 2022 Aug 22;20(1):262. doi: 10.1186/s12916-022-02460-8. PMID 35989356